CLINICAL TRIAL: NCT06514235
Title: EMBRAVE: IntErnational Observational Study on Primary Chemoradiotherapy and iMage-based Adaptive BRAchytherapy for Vaginal cancEr
Brief Title: Image-guided Brachytherapy for Vaginal Cancer (EMBRAVE)
Acronym: EMBRAVE
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Aarhus University Hospital (Other); Amsterdam University Medical Center (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Pitié-Salpêtrière Hospital (Other); Leiden University Medical Center (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Remi A. Nout, Prof. dr., Erasmus Medical Center
Other Study IDs: MEC-2021-0820; PaNaMa ID 6517 (Other: ErasmusMC)
Record Dates: First submitted 2024-07-04; First posted 2024-07-23 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Vaginal Neoplasms
MeSH Terms: conditions — Vaginal Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary vaginal cancer and Vaginal recurrence from any gynaecological cancer: Adult patients with vaginal cancer treated with curative intent by primary radio(chemo)therapy and MRI based image-guided adaptive brachytherapy according to the protocol target concept.
  Interventions: Other: Observational study (Non-interventional study)

INTERVENTIONS:
Other: Observational study (Non-interventional study) — This is an observational study.

SUMMARY:
The goal of this clinical study is to improve clinical outcomes of patients with vaginal cancer including vaginal recurrences who are treated with curative intent by primary radio(chemo)therapy and image-guided adaptive brachytherapy (IGABT).

Being an observational, prospective registration study, wherein neither an experimental treatment is compared to the standard treatment, nor groups of patients are compared.

The specific aims are:

* to develop evidence-based recommendations for curative intent treatment with primary radio(chemo)therapy and IGABT.
* to identify prognostic parameters for oncological outcomes, morbidity and quality of life.

The study aims to enroll at least 300 patients. Oncological events will be evaluated at 2 and 5 years of follow-up. Acute and late morbidity events will be evaluated at end of treatment, 2 and 5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

o Histologically proven primary vaginal cancer, vaginal carcinoma in situ (VAIN) or vaginal recurrence, per WHO classification.

Histological proven stage I-IVA primary vaginal cancer: squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the vagina, other epithelial carcinoma's and carcinoma in situ

* Histological proven vaginal recurrence from any gynaecological cancer for whom curative treatment is envisioned that includes image guided adaptive brachytherapy according to the target concept.
* Para-aortic lymph node metastasis below L1-L2 interspace are allowed
* Macroscopic visible tumour present on MRI and/or gynaecological examination at diagnosis.
* Planned IGABT treatment with MRI-guided adaptive brachytherapy (at least the 1st fraction contouring and planning on MRI; CT for later fractions is allowed):

  * External beam radio(chemo)therapy followed by IGABT
  * IGABT alone for stage I <2cm or carcinoma in situ
* Treatment with curative intent
* Written informed consent

Exclusion Criteria:

* Primary vaginal cancers with involvement of the ostium of the cervix or vulva (these should be classified as cervical cancer or vulvar cancer, respectively)
* Metastatic disease beyond para-aortic region L1-L2 interspace
* Sarcomas and melanomas.
* Treatment only by external beam radiotherapy without brachytherapy to boost the primary disease
* Primary vaginal cancer: treatment by primary surgery or debulking surgery
* Vaginal recurrences: treatment by primary surgery or debulking surgery
* Treatment with neo-adjuvant chemotherapy followed by surgery
* Treatment with radiotherapy followed by surgery
* Previous pelvic or abdominal radiotherapy
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with primary vaginal cancer stage I-IVA or vaginal recurrence from any gynaecologial cancer who are treated with curative intent by primary radio(chemo)therapy and MRI based image-guided adaptive brachytherapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2033-11-30 (Estimated); Study Completion 2033-11-30 (Estimated)

PRIMARY OUTCOMES:
Local failure | 2 and 5 years of follow-up
  A new, recurrent or progressive residual tumor within the external beam low-risk clinical target volume (CTV-TLR).
Late physician-assessed morbidity and patient reported outcomes | 2 and 5 years of follow-up
  Physician-assessed (CTCAE v.5) and Patient Reported Outcome (EORTC C30, selected items of CX24, EN24 and VU34).
Acute physician-assessed morbidity and patient reported outcomes | End of Treatment
  Physician-assessed (CTCAE v.5) and Patient Reported Outcome (EORTC C30, selected items of CX24, EN24 and VU34).

SECONDARY OUTCOMES:
Other oncological outcomes | 2 and 5 years of follow-up
  Regional failure, distant metastasis, disease free survival, disease-specific survival, overall survival.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT06514235/Prot_SAP_001.pdf